CLINICAL TRIAL: NCT07011706
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ATI-045 in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: ATI-045 Versus Placebo in Patients With Moderate-to-Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-045-AD-201
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Atopic; Dermatitis; AD; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-045 group (Experimental): ATI-045 group
  Interventions: Drug: ATI-045
- Placebo group (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATI-045 — ATI-045 group
  Arms: ATI-045 group
Drug: Placebo — Placebo group
  Arms: Placebo group

SUMMARY:
This study evaluates ATI-045 versus placebo in patients with Moderate-to-Severe Atopic Dermatitis.

DETAILED DESCRIPTION:
A Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ATI-045 in Patients with Moderate-to-Severe Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic atopic dermatitis that has been present for ≥ 6 months before the screening visit and with no significant AD flares during the past 4 weeks before screening
* Have active moderate to severe AD at screening and baseline visits
* EASI score ≥ 16 and ≥10% BSA at the screening and baseline visits
* History of inadequate response to treatment for AD with topical medications; or determination that topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks)
* Patient applied a stable dose of non-medicated topical moisturizer (ideally once or twice daily) for ≥ 7 days prior to the baseline visit and agrees to continue use during study

Exclusion Criteria:

* Treatment with any of the following:

  1. Intravenous immunoglobulin within 12 weeks prior to the baseline visit (W0D1)
  2. Systemic antibiotics within 2 weeks prior to the baseline visit (W0D1)
  3. Topical antibiotics within 1 week prior the baseline visit (W0D1)
  4. Topical medicated treatment that could affect atopic dermatitis should be prohibited for at least 2 weeks prior to baseline visit. Example: topical corticosteroids, crisaborole, calcineurin inhibitors, ruxolitinib, roflumilast, tars, antimicrobials, medical devices, and bleach baths.
  5. Topical products containing urea within 1 week prior to baseline visit (W0D1)
  6. Doxepin, hydroxyzine, or diphenhydramine within 1 week prior to the baseline visit (W0D1)
  7. Patient has used systemic treatments (other than biologics) that could affect AD less than 4 weeks or 5 half-lives (whichever is longer) prior to the baseline visit (W0D1), including, but not limited to, retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine, oral/injectable corticosteroids, baricitinib, upadacitinib, and abrocitinib.
  8. Biologics for AD treatments (such as dupilumab, tralokinumab, lebrikizumab, investigational biologics) within 5 half- lives or 12 weeks, whichever is longer prior to the baseline visit (W0D1)
  9. An investigational drug (non-biologic) within 4 weeks or within 5 half-lives (if known), whichever is longer prior to the baseline visit (W0D1)
  10. Phototherapy and photochemotherapy for AD within 4 weeks prior to the baseline visit (W0D1)
  11. A live (attenuated) vaccine within 12 weeks prior to the baseline visit (W0D1)
* History of anaphylaxis following biologic therapy.
* History of allergy to corticosteroids, diphenhydramine, hydroxyzine, cetirizine, or fexofenadine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Eczema Area and Severity Index (EASI) | Baseline to Week 24
  Percent change from baseline in EASI score at Week 24

SECONDARY OUTCOMES:
Investigator Global Assessment (vIGA) treatment success (IGA-TS) | Baseline to Week 24
  Proportion of patients with validated Investigator Global Assessment (vIGA) treatment success (IGA-TS)
EASI reduction | Baseline to Week 24
  Proportion of patients with EASI reduction of 75% (EASI75), 50% (EASI50), 90% (EASI90)
Peak Pruritus Numerical Rating Scale (PP-NRS) score | Baseline to Week 24
  Change and percent change from baseline in weekly average of the daily Peak Pruritus Numerical Rating Scale (PP-NRS) score
PP-NRS improvement | Baseline to Week 24
  Proportion of patients with a 4-point improvement or greater from baseline in weekly average of the daily Peak Pruritus Numerical Rating Scale (PP-NRS)
Body Surface Area (BSA) | Baseline to Week 24
  Change from baseline in BSA
Incidence and severity of safety measurements | From Baseline to Week 34
  Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) after first study drug dose on W0D1 until patient's last visit.
Anti-ATI-045 antidrug antibody (ADA) | From Baseline to Week 34
  ADA evaluation

CONTACTS AND LOCATIONS:
Locations (56):
- United States (49):
  - Aclaris Clinical Site, Phoenix, Arizona
  - Aclaris Clinical Site, Tucson, Arizona
  - Aclaris Study Site, Bryant, Arkansas
  - Aclaris Clinical Site, Beverly Hills, California
  - Aclaris Study Site, Encinitas, California
  - Aclaris Clinical Site, Encino, California
  - Aclaris Clinical Site, Huntington Beach, California
  - Aclaris Study Site, Los Angeles, California
  - Aclaris Study Site, Oceanside, California
  - Aclaris Study Site, Santa Monica, California
  - Aclaris Clinical Site, Sherman Oaks, California
  - Aclaris Clinical Site, Thousand Oaks, California
  - Aclaris Study Site, Coral Gables, Florida
  - Aclaris Clinical Site, Hollywood, Florida
  - Aclaris Clinical Site, Jacksonville, Florida
  - Aclaris Clinical Site, Margate, Florida
  - Aclaris Study Site, North Miami Beach, Florida
  - Aclaris Study Site, Sweetwater, Florida
  - Aclaris Study Site, Tampa, Florida
  - Aclaris Clinical Site, Wellington, Florida
  - Aclaris Clinical Site, Atlanta, Georgia
  - Aclaris Clinical Site, Savannah, Georgia
  - Aclaris Study Site, Boise, Idaho
  - Aclaris Study Site, Clarksville, Indiana
  - Aclaris Study Site, Indianapolis, Indiana
  - Aclaris Clinical Site, Lafayette, Indiana
  - Aclaris Study Site, Bowling Green, Kentucky
  - Aclaris Clinical Site, Ann Arbor, Michigan
  - Aclaris Study Site, Auburn Hills, Michigan
  - Aclaris Clinical Site, Troy, Michigan
  - Aclaris Clinical Site, Ridgeland, Mississippi
  - Aclaris Study Site, Saint Joseph, Missouri
  - Aclaris Clinical Site, Missoula, Montana
  - Aclaris Study Site, New York, New York
  - Aclaris Clinical Site, New York, New York
  - Aclaris Clinical Site, The Bronx, New York
  - Aclaris Clinical Site, Cary, North Carolina
  - Aclaris Clinical Site, Wilmington, North Carolina
  - Aclaris Study Site, Camp Hill, Pennsylvania
  - Aclaris Clinical Site, Philadelphia, Pennsylvania
  - Aclaris Clinical Site, Myrtle Beach, South Carolina
  - Aclaris Clinical Site, Dallas, Texas
  - Aclaris Clinical Site, Houston, Texas
  - Aclaris Study Site, San Antonio, Texas
  - Aclaris Clinical Site, The Woodlands, Texas
  - Aclaris Clinical Site, Providence, Utah
  - Aclaris Study Site, Norfolk, Virginia
  - Aclaris Clinical Site, Seattle, Washington
  - Aclaris Clinical Site, Spokane, Washington
- Canada (7):
  - Aclaris Clinical Site, Barrie, Ontario
  - Aclaris Site, Markham, Ontario
  - Aclaris Site, Mississauga, Ontario
  - Aclaris Site, Richmond Hill, Ontario
  - Aclaris Clinical Site, Toronto, Ontario
  - Aclaris Site, Toronto, Ontario
  - Aclaris Clinical Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No